CLINICAL TRIAL: NCT01623505
Title: Interventions for Cardiovascular Disease: "Real-World" Effectiveness of Combined Pharmacotherapy and Behavioural Counseling for Smoking Cessation
Brief Title: Reducing Cardiovascular Disease by Combining Smoking Cessation Pharmacotherapy and Behavioural Counseling
Acronym: RW
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other)
Responsible Party: Principal Investigator, Heather Tulloch, Principal Investigator, Ottawa Heart Institute Research Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HIPRC-6614
Record Dates: First submitted 2011-07-13; First posted 2012-06-20 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Smoking Cessation; Psychiatric Illness
Keywords: Smoking Cessation; Psychiatric Illness; Pharmacotherapy
MeSH Terms: conditions — Smoking Cessation; Mental Disorders | interventions — Varenicline; Chewing Gum; Nebulizers and Vaporizers; Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Champix (Experimental)
  Interventions: Drug: Champix
- Long & Combination patch treatment (Experimental)
  Interventions: Drug: Transdermal Nicoderm patch combined with gum or inhaler
- Standard patch treatment (Experimental)
  Interventions: Drug: Transdermal Nicoderm patch

INTERVENTIONS:
Drug: Champix — Participants receiving this treatment will start the medication on the day of the baseline assessment and set a target quit date within the 8 to 14 day period after baseline. Participants in this group will receive a 12-week supply of varenicline. Treatment will begin 2 weeks before the target quit date and continue for 10 weeks after the target quit date. Participants will be prescribed 0.5 mg once daily for 3 days, 0.5 mg twice daily for 4 days, and 1 mg twice daily for 11 weeks. Participants will be given the option of extending their treatment to a maximum of up to 24 weeks of varenicline.
  All participants will receive six 15-minute counselling sessions from a nurse-counsellor specializing in smoking cessation.
  Other Names: Chantix
  Arms: Champix
Drug: Transdermal Nicoderm patch combined with gum or inhaler — Participants receiving this treatment will set a quit date within 2 weeks after baseline assessment and apply the patch on that day. This group will follow the same regimen as the "standard patch treatment", but is not limited to a fixed dosing strategy. Participants will be advised on the titration of patch (increase or decrease in dosage) to ensure elimination of withdrawal symptoms (maximum dosage of 35mg/day, maximum treatment of up to 22 weeks). Participants will be provided with either gum or inhaler to manage cravings.
  All participants will receive six 15-minute counselling sessions from a nurse-counsellor specializing in smoking cessation.
  *Off-label dosage approved by Health Canada via "No Objection" letter.
  Other Names: Habitrol
  Arms: Long & Combination patch treatment
Drug: Transdermal Nicoderm patch — Participants receiving this treatment group (standard treatment)will set a target quit date within the 2 weeks after baseline assessment and start to apply the patch on that day. This treatment will consist of a 10-week supply of nicotine patches. The initial dosage will be determined from the average number of cigarettes smoked each day as per the manufacturer's recommendation. Participants smoking ≥ 20 cigarettes per day will be prescribed 21 mg/24 hours for 6 weeks, 14 mg/24 hours for 2 weeks, and 7 mg/24 hours for 2 weeks. Participants smoking 11 - 20 cigarettes per day will be prescribed 14 mg/24 hours for 6 weeks, and 7 mg/24 hours for 4 weeks.
  All participants will receive six 15-minute counselling sessions from a nurse-counsellor specializing in smoking cessation.
  Other Names: Habitrol
  Arms: Standard patch treatment

SUMMARY:
Research Aims

The aims of this research study are:

1. To determine which of the following three smoking cessation medications is most effective in achieving cessation:

   * Nicotine Patch
   * Nicotine Patch + gum or inhaler
   * Varenicline (Champix;
2. To investigate how often participants experience neuropsychiatric symptoms over the course of their cessation attempt and to assess whether:

   * They occur more often when taking one medication versus another
   * They occur more often in those with or without psychiatric illnesses.

Hypotheses to be Tested

The hypotheses to be tested include the following:

1. The CO-confirmed continuous abstinence rate from 5 weeks to 52 weeks following a target quit date will be significantly higher in smokers receiving long-term transdermal NRT in combination with other NRT products or those receiving varenicline compared to those receiving transdermal NRT alone.
2. Some participants will experience neuropsychiatric symptoms during their cessation attempt, and those in the varenicline group will experience a greater incidence of neuropsychiatric symptoms than those in the groups receiving transdermal NRT alone or in combination with other NRT products. Patients with psychiatric illnesses will report higher levels of withdrawal symptoms than those without psychiatric illnesses.

DETAILED DESCRIPTION:
Participants will be recruited from the UOHI Smoking Cessation Clinic and via media advertisements. Following the baseline assessment, participants will be randomly assigned to one of three groups:

1. 10-week standard regimen of transdermal NRT (NRT);
2. Long duration of transdermal NRT in combination with other NRT products (NRT+); or
3. Varenicline (VR).

Participants assigned to the "NRT" standard regimen group will follow a 10-week treatment of nicotine patches alone.

Participants assigned to the "NRT+" long-duration group will follow the same regimen as the NRT group, but will not be limited to a fixed declining dose strategy, nor limited to a 10-week duration (potential maximum dosage of 35mg/day and maximum treatment duration of up to 22 weeks). Participants will also be provided with other NRT products (i.e., gum or inhaler).

Participants assigned to the "VR" group will start the medication on the day of the baseline assessment and set a target quit date any time within the 8 to 14 day period after baseline. Participants will receive a 12-week supply of varenicline with a possible extension of up to 24 weeks.

All participants will receive six 15-minute counselling sessions from a nurse-counsellor specializing in smoking cessation in accordance with nursing best-practice guidelines. These sessions occur at 1, 3, 5, 8, and 10 weeks post target quit date. Counselling sessions will focus on practical counselling (problem solving and skills training) and social support.

During the treatment phase, participants will complete questionnaires measuring withdrawal and neuropsychiatric symptoms at 1, 3, 5, 8, and 10 weeks. These questionnaires will also be completed at 22 and 52 weeks after the target quit date.

ELIGIBILITY:
Inclusion Criteria:

* Participant is a current smoker (≥ 10 cigarettes per day in the preceding\ six months);
* Participant is willing to make a quit attempt in the 2-4 weeks after initial screening for eligibility;
* Participant is 18 years of age and older;
* Participant is willing to provide informed consent.

Exclusion Criteria:

* Participant is currently using or has used any intervention medications in the previous 6 months (i.e, Champix (varenicline); and/or Nicotine replacement therapy (patch, gum, inhaler, lozenge));
* Participant has contraindication(s) to any of the following smoking cessation medications:

  * Nicotine replacement therapy (allergic reaction to adhesive; serious cardiac arrhythmias (e.g., tachycardia); participant is during the immediate post-myocardial infarction period (i.e. incident has occurred within the last 10 days); severe or worsening angina pectoris; participant has had a recent cerebral vascular accident);
  * Varenicline (end-stage renal disease; use of cimetidine (by participants with severe renal impairment); previous allergic reaction to varenicline);
* Pregnant or breastfeeding women or those intending to become pregnant in the next year;
* Current or previous (in the last 3 months) substance abuse;
* Unable to provide informed consent due to unstable psychiatric symptoms (e.g., active, untreated psychosis or suicidality);
* Participant is unable to read and understand English or French;
* In order to prevent contamination across groups, only one person per household may participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 738 (Actual)
Dates: Start 2010-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be measured at 5, 10, 22, and 52 weeks after the target quit date and include: CO confirmed continuous abstinence from 5-10 weeks, 5-22 weeks and 5-52 weeks. | 5-10 weeks, 5-22 weeks, and 5-52 weeks post target quit date

SECONDARY OUTCOMES:
The secondary outcome will include withdrawal and neuropsychiatric symptoms (e.g., depression, anxiety, suicidal ideation, anger/aggression). These variables will be measured at 1, 3, 5, 8, 10, 22, and 52 weeks following the target quit date. | 1, 3, 5, 8, 10, 22, and 52 weeks post target quit date

CONTACTS AND LOCATIONS:
Overall Officials: Heather E Tulloch, PhD, Principal Investigator — Ottawa Heart Institute Research Corporation; Andrew Pipe, MD, Study Chair — Ottawa Heart Institute Research Corporation; Robert Reid, MBA PhD, Study Chair — Ottawa Heart Institute Research Corporation; Charl Els, MD, Study Chair — University of Alberta
Locations (1):
- University of Ottawa Heart Insitute - Prevention and Wellness Centre, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Aubin HJ, Bobak A, Britton JR, Oncken C, Billing CB Jr, Gong J, Williams KE, Reeves KR. Varenicline versus transdermal nicotine patch for smoking cessation: results from a randomised open-label trial. Thorax. 2008 Aug;63(8):717-24. doi: 10.1136/thx.2007.090647. Epub 2008 Feb 8. PMID 18263663
- [Background] Gonzales D, Rennard SI, Nides M, Oncken C, Azoulay S, Billing CB, Watsky EJ, Gong J, Williams KE, Reeves KR; Varenicline Phase 3 Study Group. Varenicline, an alpha4beta2 nicotinic acetylcholine receptor partial agonist, vs sustained-release bupropion and placebo for smoking cessation: a randomized controlled trial. JAMA. 2006 Jul 5;296(1):47-55. doi: 10.1001/jama.296.1.47. PMID 16820546
- [Background] Hughes JR, Keely J, Naud S. Shape of the relapse curve and long-term abstinence among untreated smokers. Addiction. 2004 Jan;99(1):29-38. doi: 10.1111/j.1360-0443.2004.00540.x. PMID 14678060
- [Background] Clinical Practice Guideline Treating Tobacco Use and Dependence 2008 Update Panel, Liaisons, and Staff. A clinical practice guideline for treating tobacco use and dependence: 2008 update. A U.S. Public Health Service report. Am J Prev Med. 2008 Aug;35(2):158-76. doi: 10.1016/j.amepre.2008.04.009. PMID 18617085
- [Background] Stapleton JA, Watson L, Spirling LI, Smith R, Milbrandt A, Ratcliffe M, Sutherland G. Varenicline in the routine treatment of tobacco dependence: a pre-post comparison with nicotine replacement therapy and an evaluation in those with mental illness. Addiction. 2008 Jan;103(1):146-54. doi: 10.1111/j.1360-0443.2007.02083.x. Epub 2007 Nov 19. PMID 18028247
- [Background] Lasser K, Boyd JW, Woolhandler S, Himmelstein DU, McCormick D, Bor DH. Smoking and mental illness: A population-based prevalence study. JAMA. 2000 Nov 22-29;284(20):2606-10. doi: 10.1001/jama.284.20.2606. PMID 11086367
- [Background] Warner KE, Burns DM. Hardening and the hard-core smoker: concepts, evidence, and implications. Nicotine Tob Res. 2003 Feb;5(1):37-48. doi: 10.1080/1462220021000060428. PMID 12745505
- [Background] Grant BF, Hasin DS, Chou SP, Stinson FS, Dawson DA. Nicotine dependence and psychiatric disorders in the United States: results from the national epidemiologic survey on alcohol and related conditions. Arch Gen Psychiatry. 2004 Nov;61(11):1107-15. doi: 10.1001/archpsyc.61.11.1107. PMID 15520358
- [Background] Slovinec D'Angelo ME, Reid RD, Hotz S, Irvine J, Segal RJ, Blanchard CM, Pipe A. Is stress management training a useful addition to physician advice and nicotine replacement therapy during smoking cessation in women? Results of a randomized trial. Am J Health Promot. 2005 Nov-Dec;20(2):127-34. doi: 10.4278/0890-1171-20.2.127. PMID 16295704
- [Derived] Theodoulou A, Chepkin SC, Ye W, Fanshawe TR, Bullen C, Hartmann-Boyce J, Livingstone-Banks J, Hajizadeh A, Lindson N. Different doses, durations and modes of delivery of nicotine replacement therapy for smoking cessation. Cochrane Database Syst Rev. 2023 Jun 19;6(6):CD013308. doi: 10.1002/14651858.CD013308.pub2. PMID 37335995
- [Derived] Tulloch HE, Pipe AL, Els C, Clyde MJ, Reid RD. Flexible, dual-form nicotine replacement therapy or varenicline in comparison with nicotine patch for smoking cessation: a randomized controlled trial. BMC Med. 2016 Jun 7;14:80. doi: 10.1186/s12916-016-0626-2. PMID 27233840
- [Derived] Tulloch HE, Pipe AL, Clyde MJ, Reid RD, Els C. The Quit Experience and Concerns of Smokers With Psychiatric Illness. Am J Prev Med. 2016 Jun;50(6):709-718. doi: 10.1016/j.amepre.2015.11.006. Epub 2015 Dec 17. PMID 26711162